CLINICAL TRIAL: NCT02855034
Title: Evaluation of Discriminating Power of Two Biomarkers (Protein S100B/Copeptin) in the Evaluation of Cerebral Lesions Due to Head Injuries in Infants and Children
Brief Title: Evaluation of Discriminating Power of Two Biomarkers in the Evaluation of Cerebral Lesions Due to Head Injuries in Infants and Children
Acronym: TCOP100
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruiting control patients to the emergency department
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9546; 2015-A00553-46 (Other: Agence Nationale de Sécurité des Médicaments)
Record Dates: First submitted 2016-08-01; First posted 2016-08-04 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Traumatic Brain Injury
Keywords: child and infant; Blood samples
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood sample (Other): All the patients performed the same blood samples for dosage: copeptin, S-100B, GFAP, NFL and UCHL-1 proteins
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Blood samples for dosage: copeptin and protein S100B

SUMMARY:
Head injury is a frequent motive of consultation in paediatric emergency units and the first cause of mortality in infants of more than one year old in developped countries. The indication of performing cerebral CT scans currently depends on clinical decision based on recommendations used in adults. In this way, 60 to 90% of scans are normal in children with head injury. CT scan is expensive and irradiating with the risk of increasing the cancer in children. Protein S100B and copeptin are biomarkers which have shown their ability to detect cerebral lesion in children with head injury. (protein S100B and /or in adults protein S100B and copetin).

It is the first clinical biological evaluation of severity of head injury based on dosing of copeptin alone or associated with protein S100B.

Furthermore, the evaluation of the biomarkers GFAP, NFL, Tau and UCH-L1 is today necessary from a scientific point of view and to optimize the diagnostic and prognostic value of these biomarkers which can be combined. Indeed, these protein biomarkers are biologically linked to the protein S100B and copeptin, and will allow a more specific and more thorough evaluation of the presence of brain damage at the cellular level. More specifically, the measurement of the S-100B and GFAP proteins will allow evaluation of gliovascular damage while those of copeptin, NFL, Tau and UCH-L1 proteins will allow evaluation of neuronal damage. The assay of these different biomarkers will also be carried out on a control population, without head injury or neurological or inflammatory pathologies, in order to establish the standards of these biomarkers on a pediatric population of similar age.

DETAILED DESCRIPTION:
265 children or infants will be recruited during 84 months. 220 patients with a suspicion of head injury and 45 patients without head injury.

Each patient will attend a visit of inclusion and a blood sample. Just patients with a suspicion of head injury have a visit at 96 hours +/- 24 hours after the inclusion: this visit is made by phone. The patient and his parents will have to answer to a phone questionnaire

ELIGIBILITY:
Inclusion criteria for the Target Population:

* Paediatric patients aged 3 months up to 15 years
* Cranial trauma with indication of brain scanner according to risk of clinically important traumatic brain injury (high or intermediate risk), according the clinical prediction rule Pediatric Emergency Care Applied Research Network (PECARN)
* Period of 6 hours of less after cranial trauma
* Informed and written consent from one of the parents or legal representatives
* Patient must be covered by a french social security scheme

Inclusion criteria for the Control Population:

* Paediatric patients aged 3 months up to 15 years admitted to the emergency room for whom a blood sample is required
* Informed and written consent from one of the parents or legal representatives
* Patient must be covered by a french social security scheme

Exclusion criteria for the Target Population:

* A pre-existing intracranial injury or malformation, or osteogenesis imperfecta
* Coagulation disorder
* Multiple accidental trauma
* Evocative elements of mistreatment

Exclusion criteria for the Control Population:

* Cranial trauma ou suspicion of cranial trauma
* brain pathology including migraines
* Febrile syndrome
* Chronic inflammatory pathology
* Known bleeding disorder
* Evocative elements of mistreatment

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 167 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Copeptin dosage | At the inclusion
  Dosage of copeptin to determine the copeptin's performance in diagnostic of traumatic brain injury

SECONDARY OUTCOMES:
S100B protein dosage | At the inclusion
  Dosage of protein S100B to determine this protein's performance in diagnostic of traumatic brain injury
GFAP protein dosage | At the inclusion
  Dosage of GFAP protein to determine this protein's performance in diagnostic of traumatic brain injury
NFL protein dosage | At the inclusion
  Dosage of NFL protein to determine this protein's performance in diagnostic of traumatic brain injury
Tau dosage | At the inclusion
  Dosage of Tau protein to determine this protein's performance in diagnostic of traumatic brain injury
UCH-L1 dosage | At the inclusion
  Dosage of UCH-L1 protein to determine this protein's performance in diagnostic of traumatic brain injury
Combinaison of Copeptine, PS-100B, GFAP, Tau and UCH-L1 protein dosage | At the inclusion
  Combination of these biomarkers to improve early discrimination of patients with brain injury secondary to CT.

CONTACTS AND LOCATIONS:
Overall Officials: Gaëlle TOURNIAIRE, MD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babcock L, Byczkowski T, Mookerjee S, Bazarian JJ. Ability of S100B to predict severity and cranial CT results in children with TBI. Brain Inj. 2012;26(11):1372-80. doi: 10.3109/02699052.2012.694565. Epub 2012 Jun 22. PMID 22725661
- [Background] Beaudeux JL, Laribi S. [S100B protein serum level as a biomarker of minor head injury]. Ann Biol Clin (Paris). 2013 Nov;71:71-8. doi: 10.1684/abc.2013.0901. French. PMID 24235330
- [Background] Bechtel K, Frasure S, Marshall C, Dziura J, Simpson C. Relationship of serum S100B levels and intracranial injury in children with closed head trauma. Pediatrics. 2009 Oct;124(4):e697-704. doi: 10.1542/peds.2008-1493. Epub 2009 Sep 28. PMID 19786430
- [Background] Bouvier D. [Interest of S100B protein blood level determination in severe or moderate head injury]. Ann Biol Clin (Paris). 2013 Mar-Apr;71(2):145-50. doi: 10.1684/abc.2013.0812. French. PMID 23587577
- [Background] Bouvier D, Fournier M, Dauphin JB, Amat F, Ughetto S, Labbe A, Sapin V. Serum S100B determination in the management of pediatric mild traumatic brain injury. Clin Chem. 2012 Jul;58(7):1116-22. doi: 10.1373/clinchem.2011.180828. Epub 2012 Apr 23. PMID 22529109
- [Background] Janigro D, Bailey DM, Lehmann S, Badaut J, O'Flynn R, Hirtz C, Marchi N. Peripheral Blood and Salivary Biomarkers of Blood-Brain Barrier Permeability and Neuronal Damage: Clinical and Applied Concepts. Front Neurol. 2021 Feb 4;11:577312. doi: 10.3389/fneur.2020.577312. eCollection 2020. PMID 33613412
- [Background] Lin C, Wang N, Shen ZP, Zhao ZY. Plasma copeptin concentration and outcome after pediatric traumatic brain injury. Peptides. 2013 Apr;42:43-7. doi: 10.1016/j.peptides.2013.01.015. Epub 2013 Feb 8. PMID 23402790
- [Background] Mathews JD, Forsythe AV, Brady Z, Butler MW, Goergen SK, Byrnes GB, Giles GG, Wallace AB, Anderson PR, Guiver TA, McGale P, Cain TM, Dowty JG, Bickerstaffe AC, Darby SC. Cancer risk in 680,000 people exposed to computed tomography scans in childhood or adolescence: data linkage study of 11 million Australians. BMJ. 2013 May 21;346:f2360. doi: 10.1136/bmj.f2360. PMID 23694687
- [Background] Mihindu E, Bhullar I, Tepas J, Kerwin A. Computed tomography of the head in children with mild traumatic brain injury. Am Surg. 2014 Sep;80(9):841-3. PMID 25197865
- [Background] Pearce MS, Salotti JA, Little MP, McHugh K, Lee C, Kim KP, Howe NL, Ronckers CM, Rajaraman P, Sir Craft AW, Parker L, Berrington de Gonzalez A. Radiation exposure from CT scans in childhood and subsequent risk of leukaemia and brain tumours: a retrospective cohort study. Lancet. 2012 Aug 4;380(9840):499-505. doi: 10.1016/S0140-6736(12)60815-0. Epub 2012 Jun 7. PMID 22681860
- [Background] Segui-Gomez M, MacKenzie EJ. Measuring the public health impact of injuries. Epidemiol Rev. 2003;25:3-19. doi: 10.1093/epirev/mxg007. No abstract available. PMID 12923986
- [Background] Yang DB, Yu WH, Dong XQ, Du Q, Shen YF, Zhang ZY, Zhu Q, Che ZH, Liu QJ, Wang H, Jiang L, Du YF. Plasma copeptin level predicts acute traumatic coagulopathy and progressive hemorrhagic injury after traumatic brain injury. Peptides. 2014 Aug;58:26-9. doi: 10.1016/j.peptides.2014.05.015. Epub 2014 Jun 4. PMID 24905622
- [Background] Yu GF, Huang Q, Dai WM, Jie YQ, Fan XF, Wu A, Lv Y, Li YP, Yan XJ. Prognostic value of copeptin: one-year outcome in patients with traumatic brain injury. Peptides. 2012 Jan;33(1):164-9. doi: 10.1016/j.peptides.2011.11.017. Epub 2011 Nov 26. PMID 22138140
- [Background] Zhang ZY, Zhang LX, Dong XQ, Yu WH, Du Q, Yang DB, Shen YF, Wang H, Zhu Q, Che ZH, Liu QJ, Jiang L, Du YF. Comparison of the performances of copeptin and multiple biomarkers in long-term prognosis of severe traumatic brain injury. Peptides. 2014 Oct;60:13-7. doi: 10.1016/j.peptides.2014.07.016. Epub 2014 Jul 27. PMID 25076464
- See also: US Department of Health and Human Services. Center for Disease Control and Prevention. Traumatic brain injury in the United States : Emergency department visits, hospitalizations and deaths 2002-2006. — https://www.cdc.gov/traumatic-brain-injury/